CLINICAL TRIAL: NCT04524468
Title: The Impact of Different Dialysis Modalities on Right Ventricular Function in End-stage Renal Disease Patients
Brief Title: Right Ventricular Function in End-stage Renal Disease Patients
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Ersan Demirci, Principal investigator, Antalya Training and Research Hospital
Other Study IDs: 2019-398
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Transthoracic Echocardiography; Hemodialysis
Keywords: echocardiography; hemodialysis; peritoneal dialysis; right ventricle
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemodialysis patients: end-stage renal disease patients on hemodialysis
  Interventions: Diagnostic Test: Transthoracic echocardiography
- peritoneal dialysis patients: end-stage renal disease patients on peritoneal dialysis
  Interventions: Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Conventional 2-D transthoracic echocardiography was performed to all patients

SUMMARY:
Right ventricular (RV) dysfunction is a major cause of heart failure and mortality in end-stage renal disease (ESRD) patients. The aim of the study was to evaluate the long-term impacts of different dialysis modalities on RV function assessed by conventional echocardiography in ESRD patients with preserved left ventricular function. The study included 83 ESRD patients grouped as follows: peritoneal dialysis (PD; n=46) and hemodialysis with brachial arterio-venous fistula (HD; n=37). Conventional echocardiography including 2D and tissue Doppler imaging was performed in all patients. Echocardiographic parameters were compared between groups.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are the main causes of death in patients undergoing dialysis. Right ventricular (RV) dysfunction is one of the major predictors of mortality and heart failure in this patient group. It has been shown that patients undergoing hemodialysis (HD) which is usually carried out via a surgically created arteriovenous fistula (AVF) have an increased risk for pulmonary hypertension and poorer right ventricular function compared with healthy controls . However, there are few data comparing the patients undergoing HD and peritoneal dialysis (PD), in terms of echocardiographic right ventricular function.

The aim of the present study was to elucidate the impact of both long term PD and HD therapy via brachial AVF on RV function in patients with preserved left ventricular (LV) function.

Patients undergoing dialysis were grouped as follows: 46 patients on PD and 37 patients on HD with brachial AVF. All of the study patients underwent transthoracic echocardiography. Left and right ventricular parameters were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients on a regular dialysis program
* Being on dialysis at least 6 months
* >18 years old

Exclusion Criteria:

* Ischemic heart disease
* Left ventricular systolic dysfunction with an ejection fraction (EF) of less than 55 %
* Valvulopathy
* Left bundle branch block
* Atrial fibrilation
* Previous renal transplantation
* Chronic obstructive pulmonary disease
* Interstitial lung diseases
* Connective tissue disorders
* Chronic thromboembolic disease
* Congenital left-to-right shunt
* Primary pulmonary hypertension

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients on a regular dialysis program at least 6 months
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Estimation of right ventricular function in end-stage renal disease patients | 1 week
  Transthoracic echocardiography was performed to end-stage renal disease patients on hemodialysis and peritoneal dialysis for at least 6 months. Tricuspid annular plane systolic excursion (TAPSE), right ventricular fractional area change (RV FAC), Right ventricular myocardial performance index (RV MPI) and right ventricular lateral peak annular systolic velocity (Sa) were measured to estimate right ventricular function.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Ersan Demirci, MD, Principal Investigator — Antalya Research and Training Hospital
Locations (1):
- Antalya Research and Training Hospital, Antalya, Turkey (Türkiye)